CLINICAL TRIAL: NCT06224166
Title: Analysis of HPV and Biomarkers Present in the Biological Fluids of Patients Suffering From Head and Neck Cancer as a Non-invasive Strategy for Detecting Recurrence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: University of Milan (Other); Istituti Tumori Giovanni Paolo II (Network)
Responsible Party: Sponsor
Other Study IDs: RS1826/23
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Head and Neck Tumors
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — tissue samples, blood and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Collection and use of tissue samples, blood and saliva — For tissue collection, tumor and surrounding tissues will be used healthy specimens taken during surgical removal, according to clinical practice. Blood and saliva sampling will be carried out at different times:
  i) the day before surgery; ii) the day after surgery (only for blood); iii) at the time of patient discharge (approximately 15 days after surgery); iii) during the check-up visit scheduled to monitor the follow-up (FU)

SUMMARY:
Multicenter, non-interventional, retrospective/prospective biological study on patients affected by head and neck tumors, for which the collection and use of tissue samples, blood and saliva for the detection of HPV-DNA/RNA and miRNA.

DETAILED DESCRIPTION:
For each patient they will come collected tissue, blood and saliva samples. In particular, as regards tissue collection, tumor and neighboring tissues will be used healthy specimens taken during surgical removal, according to clinical practice.

The fresh tissues thus collected will be stored in RNA-later before freezing at - 80°C.

Furthermore, blood and saliva samples will be taken at different times, in particular:

i) the day before surgery; ii) the day after surgery (only for blood); iii) at the time of patient discharge (approximately 15 days after surgery); iii) during the check-up visit scheduled to monitor the patient's follow-up (FU): every 3 months for the first 2 years and every 6 months for the following 3 years.

The samples will then be used to carry out nucleic acid extraction, the DNA will instead be used to detect the presence of HPV.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Patients suffering from squamous cell tumors of the oral cavity, pharynx or larynx
* Surgical patients with HNSCC primary tumors, who have not had previous tumors in other sites or adjuvant treatments prior to surgery.
* Availability of material (tissue) and follow-up data for at least one year (retrospective part)
* Written informed consent (prospective part/patients in follow-up

Exclusion Criteria:

* Presence of distant metastases at the time of diagnosis
* Previous head and neck cancer+
* Second cancer under treatment or follow-up for less than 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from head and neck tumors, recruited in a manner consecutive among those who underwent surgery at the ENT UOC of the IRE between January 2019 and December 2021 and for which, at the start of the study, archive samples as well as i follow-up data up to at least one year after surgery. The biological samples of the cohort selected include both fresh tissue and liquid biopsy (blood and saliva) samples.
Sampling Method: Non-Probability Sample
Enrollment: 283 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-01-17 (Estimated); Study Completion 2025-01-17 (Estimated)

PRIMARY OUTCOMES:
Identification of biomarkers | 24 months
  The samples that will be collected in this study will be used to carry out nucleic acid extraction.
  In particular, the extraction of RNA and DNA from tissue samples will be carried out using the "All prep RNA/DNA miRNA universal kit" kit (Qiagen), while from blood and saliva samples it will be carried out respectively through the use of the "DNAeasy blood and tissue kit" (Qiagen) and the "Magmax Total RNA extraction kit" (Thermofisher), following the instructions given in the relevant protocol.
  The expression of tissue and circulating microRNAs will be evaluated by qRT-PCR analysis using the Taqman method (Life Technology), digital-PCR (dPCR) and Luminex platform (the latter at the IRCSS G Paolo II Tumor Institute of Bari). In particular, the use of dPCR will be necessary for those low-abundance circulating miRNAs which, with the qRT-PCR methodology, are not detectable.

SECONDARY OUTCOMES:
Evaluate HPV-DNA expression as biomarkers. | 24 months
  The DNA will be used to detect the presence of HPV and will be analyzed using dPCR and the Luminex platform. These methods are able to absolutely quantify the number of viral genomes present in the sample and also to evaluate the physical state of the virus: episomal, integrated or mixed..
Evaluate miRNA expression as biomarkers | 24 months
  To identify the prognostic role of the 4 miRNAs in the liquid biopsy, the analysis of the expression of the same miRNAs in the tissue component, in order to evaluate their possible correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Blandino, Doctor, Principal Investigator — IRCCS "Regina Elena" National Cancer Institute
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy